CLINICAL TRIAL: NCT00216918
Title: An Open-Label Pilot Study of Atomoxetine Hydrochloride to Evaluate Neuropsychological Function in Children Ages 6 to 10 Years With Attention-Deficit/Hyperactivity Disorder.
Brief Title: Neuropsychological Functioning in Children With Attention-Deficit/Hyperactivity Disorder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9721; B4Z-CA-S013
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride

SUMMARY:
The purpose of this study is to evaluate the change in neuropsychological status from baseline to 6 months post-initiation of atomoxetine treatment in children ages 6 to 10.5 diagnosed with ADHD.

ELIGIBILITY:
A) Patients:

Inclusion Criteria:

1. Patients must have ADHD, be outpatients, who are at least 6 years of age and not more than 10 years 6 months of age at Visit 1 so that all testing will be completed before the child reaches age 11.
2. Patients must have moderately severe symptoms of ADHD.
3. Patients must be able to swallow study drug capsules.

Exclusion Criteria:

1. Patients must not have Bipolar disorder, psychosis, autism, Asperger's syndrome, pervasive developmental disorder, or seizure disorder.
2. Patients must not be home-schooled.

B) Controls:

Subjects will be recruited by the investigator, age and gender-matched to the atomoxetine-treated patients.

Inclusion Criteria:

1) Control subjects must be assessed to be not diagnosed with a psychiatric disorder or a medically significant disorder

Exclusion Criteria:

1) Subjects must not be home-schooled.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2005-09; Study Completion 2006-06

PRIMARY OUTCOMES:
The neuropsychological status in five domains as measured by the change in the NEPSY from baseline to 6 months post-initiation of atomoxetine treatment in children ages 6 to 10.5 diagnosed with ADHD.

SECONDARY OUTCOMES:
Assess changes in executive function and attention;Compare changes in neuropsychological status in a normal control group, gender and age matched to atomoxetine-treated patients at baseline and 6 months
Efficacy of atomoxetine after 2 and 6 months, or endpoint from baseline;Assess the correlation of change from baseline to 6 months, or at study discontinuation, in ADHD symptoms with change from baseline in the neuropsychological functioning
Assess the relationships of change from baseline to approximately 2 and 6 months, or endpoint in the core symptoms of ADHD with the changes in functional outcomes as assessed by the WFIRS-P
Examine the French language version of the WFIRS-P questionnaire's psychometric properties including internal consistency and responsiveness to change.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec, Canada

REFERENCES:
- [Derived] Dickson RA, Maki E, Gibbins C, Gutkin SW, Turgay A, Weiss MD. Time courses of improvement and symptom remission in children treated with atomoxetine for attention-deficit/hyperactivity disorder: analysis of Canadian open-label studies. Child Adolesc Psychiatry Ment Health. 2011 May 11;5:14. doi: 10.1186/1753-2000-5-14. PMID 21569378